CLINICAL TRIAL: NCT04560738
Title: A Phase 1, Single Center, Open Label Study to Evaluate the Metabolism and Excretion of [14C] CC 92480 in Healthy Male Subjects
Brief Title: A Study to Evaluate the Metabolism and Excretion of [14C]-CC-92480 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CC-92480-CP-004; U1111-1257-8762 (Registry Identifier: WHO)
Record Dates: First submitted 2020-09-21; First posted 2020-09-23 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; CC-92480; Healthy male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of [14C]-CC-92480 (Experimental): [14C]-CC-92480 will be administered as an oral solution. A single oral dose of [14C]-CC-92480, containing approximately 2 μCi of radioactivity, will be administered on Day 1 under fasted conditions.
  Interventions: Drug: [14C]-CC-92480

INTERVENTIONS:
Drug: [14C]-CC-92480 — Oral

SUMMARY:
This is a single-center, open-label study to be conducted in healthy adult male participants. This study is designed to characterize the biotransformation and excretion of [14C]-CC-92480 and to evaluate the safety and tolerability of [14C]-CC-92480 following a single oral dose of [14C]-CC-92480.

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy the following criteria to be enrolled in the study:

1. Participant is ≥ 18 and ≤ 55 years of age at the time of signing the informed consent form (ICF).
2. Participant is male.
3. Participant must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
4. Participant is willing and able to adhere to the study visit schedule and other protocol requirements.
5. Participant is in good health, as determined by the Investigator at the time of signing the ICF.
6. Participant agrees to abide by the requirements and restrictions outlined in the CC-92480 Pregnancy Prevention Plan for Participants in Clinical Trials.
7. Participant must practice true abstinence or agree to use a barrier method of birth control (condoms not made out of natural [animal] membrane [latex condoms are recommended]) during sexual contact with a pregnant female or a FCBP while participating in the study and for at least 90 days following administration of CC-92480, even if he has undergone a successful vasectomy. A FCBP is a female who: 1) has achieved menarche at some point; 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months).
8. Participant has a body mass index (BMI) ≥ 18 and ≤ 33 kg/m2 at the time of signing the ICF.
9. Participant has clinical laboratory safety test results, including alanine aminotransferase (ALT)/aspartate aminotransferase (AST) results, that are within normal limits or considered not clinically significant by the Investigator.

   1. Platelet count and absolute lymphocyte count (ALC) must be above the lower limit of normal at screening.
   2. Absolute neutrophil counts (ANC) must be greater than 2500/microliter.
10. Participant is afebrile, with supine systolic BP ≥ 90 and ≤ 140 mm Hg, supine diastolic BP ≥ 50 and ≤ 90 mm Hg, and pulse rate ≥ 40 and ≤ 110 bpm at screening.
11. Participant has a normal or clinically acceptable 12-lead ECG, with a QT interval corrected for heart rate using Fridericia's formula (QTcF) value ≤ 430 msec, at screening.

Exclusion Criteria:

The presence of any of the following will exclude a participant from enrollment:

1. Participant has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the participant from participating in the study.
2. Participant has a history of chronic pruritus or clinically significant chronic dermatologic disorder.
3. Participant has contraindication or intolerance to first-generation antihistamine medications.
4. Participant has a history of benign ethnic neutropenia.
5. Participant has a history of any clinically significant and relevant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies, or other major disorders as determined by the Investigator.
6. Participant has any condition, including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he were to participate in the study.
7. Participant has any condition that confounds the ability to interpret data from the study.
8. Participant was exposed to an investigational drug (new chemical entity) within 30 days prior to dosing or 5 half-lives of that investigational drug, if known (whichever is longer).
9. Participant has used any prescribed systemic or topical medication (including but not limited to analgesics, anesthetics, etc) within 14 days or 5 half-lives of that medication, whichever is longer, prior to dosing.
10. Participant has used any non-prescribed systemic or topical medication (including vitamin/mineral supplements and herbal medicines) within 7 days prior to dosing.
11. Participant has used CYP3A inducers and/or inhibitors (including St. John's Wort) within 30 days prior to dosing. The Indiana University "Cytochrome P450 Drug Interaction Table" should be utilized to determine inducers and/or inhibitors of CYP3A (http://medicine.iupui.edu/clinpharm/ddis/table.aspx).
12. Participant has any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism, and excretion, eg, bariatric procedure.

    Note: prior appendectomy is acceptable, but prior cholecystectomy would result in exclusion from the study.
13. Participant donated blood or plasma within 8 weeks prior to dosing to a blood bank or blood donation center.
14. Participant has a history of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years prior to dosing, or positive drug test reflecting consumption of illicit drugs.
15. Participant has a history of alcohol abuse (as defined by the current version of the DSM) within 2 years prior to dosing, or positive alcohol test.
16. Participant is known to have serum hepatitis or known to be a carrier of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCV Ab), or have a reactive result to the test for human immunodeficiency virus (HIV) antibodies at screening.
17. Participant has a history of smoking/use of tobacco or nicotine-containing products within 3 months prior to check-in (Day -1).
18. Participant has received immunization with a live or live-attenuated vaccine within 2 months prior to dosing or is planning to receive immunization with a live or live-attenuated vaccine for 2 months following dosing.
19. Participant participated in a radiolabeled drug study, where exposures are known to the Investigator, within the previous 4 months prior to check-in (Day -1); or participated in a radiolabeled drug study, where exposures are not known to the Investigator, within the previous 6 months prior to check-in (Day -1). The total 12-month exposure from this study and a maximum of 2 other previous studies within 4 to 12 months of this study will be within the CFR-recommended levels considered safe: less than 5000 mrem whole body annual exposure, with consideration given to the half-lives of the previous radiolabeled study drugs received.
20. Participant was exposed to significant radiation (eg, serial X-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring) within 12 months prior to check-in (Day -1).
21. History of less than 1 to 2 bowel movements per day.
22. Participant is part of the study site personnel or a family member of the study site staff.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-05-13 (Actual)

PRIMARY OUTCOMES:
Cumulative excretion of [14C]-RA | Up to approximately 15 days
  The total recovery of radioactivity (RA) will be computed as the sum of the cumulative excretion (as % dose) in urine and feces (and vomit, if applicable).
Pharmacokinetics -Tmax of total radioactivity, CC-92480 and its metabolites | Up to approximately 15 days
  Time to reach maximum total radioactivity or concentration of CC-92480 and its metabolites
Pharmacokinetics - Cmax of total radioactivity, CC-92480 and its metabolites | Up to approximately 15 days
  Maximum total radioactivity or concentration of CC-92480 and its metabolites
Pharmacokinetics - AUC0-t of total radioactivity, CC-92480 and its metabolites | Up to approximately 15 days
  Area under the concentration-time curve from time zero to the last measured time point
AUC0-inf of total radioactivity, CC-92480 and its metabolites | Up to approximately 15 days
  Area under the concentration-time curve from time zero extrapolated to infinite time
Pharmacokinetics - CL/F of total radioactivity, CC-92480 and its metabolites | Up to approximately 15 days
  Apparent oral clearance
Pharmacokinetics - Vz/F of total radioactivity, CC-92480 and its metabolites | Up to approximately 15 days
  Apparent volume of distribution
Pharmacokinetics - t1/2 of total radioactivity, CC-92480 and its metabolites | Up to approximately 15 days
  Terminal elimination half-life
Metabolic profiling in urines and feces | Up to approximately 15 days
  The percentage of the administered dose attributed to CC-92480 and its metabolites in urine and feces

SECONDARY OUTCOMES:
Adverse Events (AEs) | From enrollment until at least 28 days after completion of study treatment
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Covance Clinical Research Unit Inc, Madison, Wisconsin, United States